CLINICAL TRIAL: NCT01202734
Title: An Open-label, Single-Ascending-Dose Study to Investigate the Pharmacokinetics and Safety of CONCERTA in Healthy Japanese Adult Male Subjects
Brief Title: A Pharmacokinetics and Safety of Methylphenidate HCl in Healthy Japanese Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CR017464
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: CONCERTA; Methylphenidate HCl; Pharmacokinetic; Safety; Adult; Men; Male
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Methylphenidate

ARMS (1):
- 001 (Experimental): Methylphenidate HCl Period 1: One tablet oral 36 mg once daily single-dose on Day 1 Period 2: Three tablets oral 18 mg once daily single-dose on Day 1 Period 3: Two tablets oral 36 mg once daily single-dose on Day 1. (Each treatment period will be separated by 3-7 days)
  Interventions: Drug: Methylphenidate HCl

INTERVENTIONS:
Drug: Methylphenidate HCl — Period 1: One tablet, oral, 36 mg, once daily, single-dose on Day 1

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics and safety of 3 single doses of Methylphenidate HCl in healthy Japanese adult male volunteers.

DETAILED DESCRIPTION:
This is an open-label (name of assigned treatment is known), single-center study of the pharmacokinetics (blood levels) and safety of 3 single doses of methylphenidate HCl administered orally (by mouth) to healthy Japanese adult male volunteers. Methylphenidate HCl is a drug that is currently approved for the treatment of adults with attention-deficit/hyperactivity disorder (ADHD) in regions outside Japan, including the United States where this study will be conducted. Volunteers will participate in the study for a maximum of 42 days. Blood samples will be collected from volunteers during the study to determine the concentration of the methylphenidate HCl in the blood after dosing. Safety will be monitored throughout the study by evaluating adverse events reported, changes in clinical laboratory test results, vital signs measurements, physical examination results, and other protocol-specified safety assessments. All volunteers will receive a single oral dose of methylphenidate HCl with 240 mL (1 cup) of noncarbonated water after at least a 10-hour fast (without eating food) during 3 treatment periods as follows: Period 1, one 36-mg tablet; Period 2, three 18-mg tablets; and Period 3, two 36-mg tablets. Treatment periods will be separated by 3 to 7 days. Volunteers will continue fasting until at least 4 hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 25.0 kg/m², inclusive
* Body weight of not less than 50 kg
* Supine (lying down) blood pressure between 90 and 140 mmHg systolic, inclusive, and not higher than 90 mmHg diastolic

Exclusion Criteria:

* History of or current medical illness judged by the investigator to be clinically significant
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, within 14 days before the first dose of study drug
* History of drug or alcohol abuse within the past 5 years
* History of smoking or use of nicotine containing substances within the previous 2 months

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of total methylphenidate HCl and its major metabolite, a-phenyl-piperidine-acetic acid (PPAA) | At protocol-specified times on Day 1 through Day 3 in Treatment Periods 1, 2, and 3

SECONDARY OUTCOMES:
The number and type of treatment-emergent adverse events | Day 1 of Period 1 through Day 3 of Period 3 (approximately 23 days)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Cypress, California, United States